CLINICAL TRIAL: NCT04440397
Title: Endoplasmic Reticulum Stress and Endometriosis Releated Pain
Brief Title: Relationship Between Endoplasmic Reticulum Stress and Pain in Patients With Endometriosis
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: xbpendo
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Endometriosis; Endoplasmic Reticulum Stress; Endometriosis-related Pain
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: xbp-1 - endometriosis patients group — Patients diagnosed with endometriosis by surgery and ultrasound and whose xbp-1 level was examined

SUMMARY:
The correlation between painful symptoms (dysmenorrhea, dysparonia, dysuria, chronic pelvic pain) symptoms and endoplasmic reticulum stress was investigated in 86 patients diagnosed with endometriosis. For this, xbp-1 (x box binding protein-1) level was measured in patients. XBP-1 is an endoplasmic reticulum stress indicator and is known to be involved in pain pathogenesis.

DETAILED DESCRIPTION:
Women between the ages of 18-50 who were diagnosed with endometriosis by surgery and ultrasound, without known rheumatological or metabolic diseases were included in the study. Most of the patients are composed of newly diagnosed patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed endometriosis with ultrasound or surgery
* no metabolic diseases
* no rheumatological diseases

Exclusion Criteria:

* Immune modulator, hormonal, anti-inflammatory use history in the last 3 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women between the ages of 18-50 who were diagnosed with endometriosis by ultrasound or surgery and who did not have any rheumatological and metaboli disease were included in the study. women with drug use indicated in the last 3 months were excluded from the study.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the correlations between the results of XBP-1 levels and the stages and pain symptoms of endometriosis. | 5 months

SECONDARY OUTCOMES:
serum XBP-1levels in patients wit endometriosis | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes